CLINICAL TRIAL: NCT04841044
Title: Health Effects of Cetoleic Acid (Helseeffekter av Ketolinsyre)
Brief Title: Health Effects of Cetoleic Acid (A Randomized Double Blinded Controlled Trial)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Oslo (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Kirsten Holven, Professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: REK 176979
Record Dates: First submitted 2021-04-08; First posted 2021-04-12 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Healthy Diet
Keywords: Omega 3 fatty acids; Sustainability; Cetoleic acid; Very long monounsaturated fatty acid; Cardiovascular disease prevention; Antiinflammation
MeSH Terms: interventions — cetoleic acid

STUDY DESIGN:
Intervention Model Description: Randomized double-blinded controlled trial (Randomized 1:1, control:intervention).
  Run-in period of 3 weeks where all participants receive the control capsules.
Who Masked: Participant, Care Provider, Investigator
Masking Description: All participant, the major investigator, study coordinator and the study staff are blinded for the randomizing. The capsules and capsule containers will only be identifiable by the ID (identifying) numbers on the containers.
  Allocation of participants to the specific intervention group is carried out by a statistician and one person not involved in conducting the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention ( Cetoleic acid) (Experimental): 6x mackerel oil (cetoleic acid: 16A%, estimated: 135 mg/g (FFA)) capsules every morning for 4 weeks
  (A%= area percent)
  Interventions: Dietary Supplement: Cetoleic acid
- Control oil (Placebo Comparator): 6x capsules control oil (Control oil= mix of anchovy oil, olive oil, high-oleic sunflower oil, rapeseed oil (cetoleic acid: 0,7 A% estimated: 6 mg/g (FFA)) every morning for 4 weeks
  (A%= area percent)
  Interventions: Dietary Supplement: Control Oil

INTERVENTIONS:
Dietary Supplement: Cetoleic acid — Very long monounsaturated fatty acid ( C22:1n-11)
  Arms: Intervention ( Cetoleic acid)
Dietary Supplement: Control Oil — Control oil consisting of: mix of anchovy oil, olive oil, high-oleic sunflower oil and rapeseed oil
  Arms: Control oil

SUMMARY:
In this Randomized Controlled Trial (RCT) we want to study how supplements of cetoleic acid ( C22:n1-11) (intervention) affect the conversion of alpha-linolenic acid (ALA) to EPA (eicosapentaenoic acid) and DHA (docosahexaenoic acid) in healthy subjects, compared to supplements with a low concentration of cetoleic acid (control).

Our primary endpoints are changes in the concentration of EPA and DHA in plasma and red blood cells.

DETAILED DESCRIPTION:
This is a randomized double-blinded controlled trial ( randomized 1:1). Study population: healthy men and women 20-70 years, BMI 20-35 kg/m2.

Study design:

* 3 weeks run-in-period where all participants consume control capsules every morning.
* Randomization intervention: control (1:1). All participants consume their capsules (control or intervention) for 4 weeks.

The intervention oil consists of a fish oil high in cetoleic acid and the control oil is a mix of different oils and low in cetoleic acid.

Power calculation and sample size:

It was expected a difference of 15% in n-3 between the groups after the intervention (Østbye et al. 2019, doi:10.1017/S0007114519001478).

The level of significance was set to 5% (two-sided) and the power to 80%. A total of thirty-eight subjects were required to participate in the study, but a high dropout rate was expected (20%) and it was considered necessary to include a total of seventy (n=70) subjects (thirty-five per arm).

ELIGIBILITY:
Inclusion Criteria:

* BMI 20-35kg/m2
* opportunity to meet for 3 visits at the Department of Nutrition, University of Oslo, during the study period.

Exclusion Criteria:

* Chronic disease (liver/kidney/metabolism)
* Alcohol overconsumption (>40g/day)
* Diabetes and high fasting blood glucose
* Pregnant/ breastfeeding or planning pregnancy during the study period
* High fish intake (>3 meals/week).
* Blood donation during the study period
* Difficulty following the study protocol.
* Smoking/snuffing
* Regularly use of anti-inflammatory drugs
* Regularly use of omega-3 supplements /cod liver oil.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-27 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
EPA and DHA in plasma | 4 weeks intervention
  EPA and DHA concentration in plasma measured at baseline and and after 4 week intervention (and as a "control measurement" at the screening visit)
EPA and DHA in red blood cells | 4 weeks
  EPA and DHA concentration and omega 3 index (EPA+DHA/total fatty acids) in red blood cells measured at baseline and and after 4 week intervention (and as a "control measurement" at the screening visit)

SECONDARY OUTCOMES:
Lipid profile- Triglycerides | 4 weeks
  Plasma levels of triglycerides measured at baseline and after 4 weeks intervention (and as a "control measurement" at the screening visit)
Lipid profile- Cholesterol | 4 weeks
  Plasma levels of cholesterol (total cholesterol, LDL-cholesterol and HDL-cholesterol) measured at baseline and after 4 weeks intervention (and as a "control measurement" at the screening visit)
Lipid profile- Apolipoproteins | 4 weeks
  Plasma levels of apolipoproteins (apoB and apoA) measured at baseline and after 4 weeks intervention (and as a "control measurement" at the screening visit)
Lipid profile- Lipoproteins | 4 weeks
  Plasma levels of Lp(a) and lipoprotein subclasses measured at baseline and after 4 weeks intervention (and as a "control measurement" at the screening visit)
Inflammatory markers | 4 weeks
  The concentration of circulating levels of inflammatory markers measured at baseline and after 4 weeks intervention ( and as a "control measurement" at screening)
Gene expression | 4 weeks
  Changes in PBMC (peripheral blood mononuclear cell) gene expression profile measured at baseline and after 4 week of intervention
Pain sensitivity | 4 weeks
  Measured by cold pressure tests at baseline and after 4 week of intervention ( and as a control measurement at screening)
Resolvins | 4 weeks
  Blood levels of resolvins (omega- 3 derivates) concentrations measured at baseline and after 4 week of intervention ( and as a control measurement at screening)
Metabolome | 4 weeks
  Changes in metabolome measured at baseline and after 4 week of intervention

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oslo, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
Data will not be sheared as individual participant data, but the results will be shared on group levels. All participants information are treated deidentified